CLINICAL TRIAL: NCT01762332
Title: Validation of Medasense Non-invasive Nociception Monitor During Surgery and Postoperative Recovery.
Brief Title: Clinical Validation of Medasense Pain Response Index (PRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: Medasense003; 0326-12-RMB (Other: Rambam Health Care Campus, Haifa, Israel)
Record Dates: First submitted 2012-12-23; First posted 2013-01-07 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2015-05

CONDITIONS: Surgery; Pain
Keywords: nociception; analgesia; intraoperative monitoring
MeSH Terms: conditions — Pain; Agnosia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low opioid level (Active Comparator): Base level of remifentanil effect side concentration: 2ng/ml Stopped recruitment (May 2014)
  Interventions: Drug: Base level of remifentanil effect side concentration: 2ng/ml
- High opioid level (Active Comparator): Base level of remifentanil effect side concentration: 4ng/ml Stopped recruitment (May 2014)
  Interventions: Drug: Base level of remifentanil effect side concentration: 4ng/ml; Other: chronic beta-blocker treatment
- chronic beta-blocker treatment (Other): Patients with chronic beta-blocker treatment prior to surgery and study. Will all be allocated to the high opioid level arm without randomization.
  Continue recruitment.
  Interventions: Other: chronic beta-blocker treatment

INTERVENTIONS:
Drug: Base level of remifentanil effect side concentration: 2ng/ml — constant remifentanil level of 2ng/ml administered using Target Control Infusion pumps.
  Other Names: Ultiva
  Arms: Low opioid level
Drug: Base level of remifentanil effect side concentration: 4ng/ml — constant remifentanil level of 4ng/ml administered using Target Control Infusion pumps.
  Other Names: Ultiva
  Arms: High opioid level
Other: chronic beta-blocker treatment — Patients from the chronic beta-blocker treatment group will not be randomized, and will all be allocated to the high opioid level group.
  Arms: High opioid level; chronic beta-blocker treatment

SUMMARY:
In our previous study, NCT01631695, we proposed and clinically evaluated the Medasense pain response index, PRI, in anesthetized patients undergoing surgery. Note: the name PRI has been changed to NoL (Nociception Level) Index.

The PRI is based on a non-linear combination of several pain-related physiological parameters into a one unique index (0-100).

In this study we aim to validate the performance of the PRI by:

1. investigating the patient's PRI response to surgical painful stimuli under different levels of analgesia:

   * Investigating patient's PRI response to surgical painful stimuli under two different levels of Remifentanil Target Control Infusion (TCI) rates.
   * Investigating patient's PRI response to standardized painful stimulus (Tetanic stimulus) with and without opioids.
2. investigating the effect of beta-blockers on PRI performance in patients taking chronic beta-blocker treatment.

The study is based on recording and analyzing the subject's physiological signals, while recording painful events, medication dosing and different clinical signs.

DETAILED DESCRIPTION:
Pain is an unpleasant sensation, ranging from slight discomfort to intense suffering. Since pain is a subjective phenomenon, it has frequently defied objective, quantitative measurements. Today, in order to measure pain, subjective uni-dimensional scales are used to quantify pain. One of the most common scale used to rate a patient's pain intensity is the Numeric Pain Scale (NPS), usually scored from 0 to 100. Hitherto, those scales are based on the subjective evaluation of pain by the patient.

During anesthesia the patient cannot communicate and therefore the verbal or other report is impossible. As a consequence, due to misrepresentation of the existence or extent of pain, care providers may fail to estimate the correct measure of pain and give too much or too little medication, leading to possible complications and adverse reactions. A validated scoring system of subject's pain level, or as in the case of an anaesthetised patient, subject's nociception level, is therefore needed.

In this study the investigators intend to test and analyze the performances of Medasense pain response index, PRI, by comparing it with other standard pain related indicators (Heart Rate (HR), Heart Rate Variability (HRV), Skin Conductance, etc) before and after painful stimuli at different levels of analgesia. In addition, in order to reduce the variability between stimuli, a standardized stimulus (Tetanic ,30 sec, 100Hz, 60mA) will be given to all patients after sleep induction and before intubation, with and without administration of Fentanyl and the values of the PRI during these stimuli will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3
* Elective surgery

Exclusion Criteria:

* Pregnancy or lactation
* History of severe cardiac arrhythmias
* Abuse of alcohol or illicit drugs
* History of mental retardation, dementia, psychiatric disorders
* Allergy to any of the drugs to be used during anesthesia and recovery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Medasense's non-invasive pain monitoring index in response to painful events | at time of surgery. 1 minute before and 1 minute after painful stimuli (for instance: intubation, skin incision, trocar insertion)
  outcome measure will be assessed one minute before painful event, and will be compared to a measure taken during the painful event.
  Note: during data analysis it became aparent that these definitions cannot be met. For example: the time of various clinical stimuli cannot be identified within seconds. Also, there is no meaning to a measure taken during event. Therefore, to avoid including part of the stimulus in the pre stimulus window, we restricted analysis to the first 30 seconds of the designated 1 minute before the event (-30 to -60 seconds). Similarly, the post stimulus window start was defined 10 seconds after the event annotation and the post stimulus window enlarged to 80 seconds.

SECONDARY OUTCOMES:
Change in all pain related physiological parameters (heart rate, heart rate variability, Plethysmograph amplitude, skin conductance, etc) in response to specific painful stimuli | at time of surgery. 1 minute before and 1 minute after painful stimuli (for instance: intubation, skin incision, trocar insertion)
  Outcome measures will be assessed one minute before painful event, and will be compared to measures taken during the painful event.
  Note: same changes as in outcome 1 measure.
Change in Medasense index/pain related physiological parameters/subjective pain assessment in response to changes in the level of analgesic drugs | at time of surgery. 1 minute before and 5 minute after analgesics administration
  Outcome measures will be assessed one minute before administration of analgesic drug, and will be compared to measures taken 5 minutes after.
  Note: after fentanyl administration - same change as in outcome 1 measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Edry, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Treister R, Kliger M, Zuckerman G, Aryeh IG, Eisenberg E. Differentiating between heat pain intensities: the combined effect of multiple autonomic parameters. Pain. 2012 Sep;153(9):1807-1814. doi: 10.1016/j.pain.2012.04.008. Epub 2012 May 29. PMID 22647429
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792